CLINICAL TRIAL: NCT00192218
Title: A Phase IV Study to Evaluate the Effectiveness of Flumist (Influenza Vaccine, Live Intranasal) Vaccination in a School-Based Intervention Program
Brief Title: Study to Evaluate the Effectiveness of FluMist Vaccination in a School-Based Intervention Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert Walker, MD, MedImmune LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MI-MA004
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

ARMS (1):
- 1 (Experimental): FluMist
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — 0.5 ml of vaccine intranasally (0.25 ml in each nostril) which contains approximately 107 TCID50 of each type

SUMMARY:
To measure the effectiveness of influenza vaccination in school children by comparing, between target(i.e., children are offered FluMist) and control (i.e., children are not offered FluMist) school families.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children enrolled in the target schools.
* Written informed consent obtained from the child's parent(s) if they agree to participate.

Exclusion Criteria:

* History of severe hypersensitivity (anaphylactic response) to egg products or previous FluMist
* FluMist is licensed exclusively for use in healthy individuals age 5-49 years. Therefore children for whom annual receipt of inactivated influenza vaccine for specific medical condition(s) is recommended will not be eligible. These conditions include:
* Asthma, other chronic pulmonary diseases, kidney disease, metabolic disease, heart disease, or hemoglobinopathy
* Immunosuppression of child
* Severe immunosuppression of a household member
* Pregnancy
* Past history of Guillian-Barre Syndrome
* Aspirin therapy within 1 month prior to FluMist or the anticipated use of aspirin containing products for one month after FluMist administration
* Administration of any inactivated vaccine within 2 weeks or any live vaccine within 4 weeks prior to receipt of FluMist
* Received anti-influenza medication in the past 48 hours
* Fever in the past 72 hours
* Moderate to severe nasal congestion (inability to breathe through the nose) or acute phase URI symptoms until the congestion has improved

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3022 (Actual)
Dates: Start 2004-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To compare the families of children in the target schools with families of children in the control schools with respect to workdays lost by adults and school days lost by children. | 7 days after each vaccination

SECONDARY OUTCOMES:
Absenteeism - To compare the families of children in the target schools to those in the control schools with respect to the overall increase in absenteeism during the influenza outbreak, using aggregated (summary) absentee rates. | between outbreak and non-outbreak weeks
Herd Community - To compare unvaccinated children in the target schools to the children in the control schools with respect to changes in absentee rates between outbreak weeks and non-outbreak weeks. | between outbreak and non-outbreak weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (2):
- United States (2):
  - Division of General Pediatrics, University of Maryland School of Medicine, Baltimore, Maryland
  - Division of Allergy and Infectious Diseases, University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Derived] King JC Jr, Stoddard JJ, Gaglani MJ, Moore KA, Magder L, McClure E, Rubin JD, Englund JA, Neuzil K. Effectiveness of school-based influenza vaccination. N Engl J Med. 2006 Dec 14;355(24):2523-32. doi: 10.1056/NEJMoa055414. PMID 17167135